CLINICAL TRIAL: NCT05522569
Title: Expanded Access Multi-Patient Experimental Treatment Involving Allogeneic Human Mesenchymal Stem Cells (Allo-hMSCs) in Subjects With Acute Ischemic Stroke (EXPAND)
Brief Title: Expanded Access Multi-Patient Experimental Treatment Involving Allogeneic Human Mesenchymal Stem Cells (hMSCs) in Subjects With Acute Ischemic Stroke (EXPAND)
Acronym: EXPAND
Status: Temporarily not available | Type: Expanded Access
Sponsor: University of Miami (Other)
Responsible Party: Principal Investigator, Dileep Raghvendra Yavagal, Professor of Clinical Medicine, University of Miami
Other Study IDs: 20201338
Record Dates: First submitted 2022-08-27; First posted 2022-08-31 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Acute Ischemic Stroke; Mesenchymal Stem Cells; Stroke, Acute; Stroke/Brain Attack; Stroke, Ischemic
Keywords: Allogeneic Mesencyhmal Stem cells; Acute Ischemic Stroke; Cell Therapy; Regenerative Therapy; Intravenous
MeSH Terms: conditions — Ischemic Stroke; Stroke

STUDY DESIGN:
Expanded Access Types: Intermediate

INTERVENTIONS:
Drug: Allogeneic human mesenchymal stem cells (Allo-hMSCs) — Participants will be treated with one intravenous (IV) infusion of 200 million allogeneic human mesenchymal stem cells (Allo-hMSCs), lasting from 40-90 minutes following an acute ischemic stroke within 9 days after stroke symptom onset.

SUMMARY:
The purpose of this study is to use an intravenous infusion of allogeneic human mesenchymal stem cells (Allo-hMSCs) to treat an acute ischemic stroke condition.

ELIGIBILITY:
Inclusion Criteria:

1. Acute ischemic stroke , had a recent (within the past 9 days), acute, cortical, hemispheric, ischemic stroke in the middle cerebral artery (MCA) distribution without a midline shift as detected by magnetic resonance imaging (MRI) as a diffusion-weighted image (DWI) abnormality
2. Qualifying Stroke Event must be confirmed by CT or MRI.
3. Age 18 to 80 years If >80 then the pre-stroke modified Rankin Score (mRS) needs to be < 1.
4. Has a National Institutes of Health Stroke Scale (NIHSS) score of 6 -15 (Right hemisphere), and 6-18 (left hemisphere) at the time of enrollment
5. Known onset time of acute symptoms
6. Subjects must have a platelet count >100,000/ Microliter(uL), hemoglobin >8gm/dl, and white blood cell count (WBC) >2,500/uL
7. Mesenchymal stem cells (MSC) infusion procedure must be performed within 9 days after stroke symptom onset
8. Is able to provide consent to participate or consent is obtained from the subject's legally authorized representative
9. Subjects who received tissue plasminogen activator (tPA) or underwent mechanical reperfusion may be included in the expanded access experimental treatment
10. Patients must be hemodynamically stable post-stroke.

Exclusion Criteria:

1. Permanent disability corresponding to a Modified Rankin Score of >1 prior to the Qualifying Stroke Event.
2. Has a medical history of neurological or orthopedic pathology with a deficit as a consequence that results in a modified Rankin Scale >1 before stroke or has a pre-existing cognitive deficit.
3. Ischemic stroke in the last 3 months, any vascular territory. Has clinically significant and/or symptomatic hemorrhage associated with stroke
4. Myocardial Infarction (MI), primary hemorrhagic or traumatic lesion of the brain within the last 3 months or identified on magnetic resonance imaging (MRI). Small hemorrhagic transformation of the acute infarct is allowed.
5. Seizure disorder
6. Developmental delay
7. Chronic kidney disease is defined as baseline serum creatinine >1.4
8. Hepatic disease or altered liver function as defined by serum glutamate pyruvate transaminase (SGPT) >150 U/L and or T. Bilirubin >1.6 mg/dL at admission
9. Pulmonary disease (e.g., chronic obstructive pulmonary disease (COPD) with oxygen requirement at rest or with ambulation, moderate to severe asthma)
10. Mechanical heart valve
11. Active malignancy or diagnosis of malignancy within 5 years prior to the start of screening or any history of chemotherapy or radiation affecting the bone marrow. Skin cancers (except for melanoma) are permitted.
12. Prior immunosuppression, including chemotherapy administration within last 3 years or current immunosuppression as defined by white blood cell count (WBC) <3 x 103 cells/ml
13. Hepatic insufficiency (bilirubin >2.5mg/dL or transaminases >5x the upper limit of normal). Patients with Gilberts syndrome are eligible for enrollment if other liver function tests are normal, regardless of bilirubin level.
14. Known HIV
15. Hemoglobin <10g/dl
16. Uncorrected coagulopathy at the time of consent defined as international normalized ratio (INR) >1.4; partial thromboplastin time (PTT) >37 sec, or thrombocytopenia (PLT<100,000)
17. Any hemodynamic instability at the time of consent (e.g., requiring continuous fluid resuscitation or ionotropic support).
18. Hypoxemia (SaO2<90%) at the time of consent, respiratory distress or persistent hypoxemia defined as SaO2 <94% for >30 minutes occurring at any time from hospital admission to time of consent. Intubation alone is not an exclusion.
19. Pregnancy or positive human chorionic gonadotropin (HCG) or lactating women
20. Subjects participating in another interventional clinical trial of an investigational therapy within 30 days of screening
21. Unable to return for follow-up visits for clinical evaluation, laboratory studies, or imaging evaluation
22. Multiple anti-platelet medications (Aggrenox is considered a single platelet agent)
23. Unable to undergo MRI or CT scan
24. Any other condition that the investigator feels would pose a significant hazard to the patient if enrolled.
25. Exclude infarct lesion size >145cc unless the NIHSS 1a remains < 1 and there is no evidence of infarct expansion or edema formation on any imaging obtained from admission up to the point just prior to infusion.
26. Exclude Intra Arterial (IA) therapy use or if there is a planned or anticipated hemicraniectomy. Diagnostic angiograms are allowed
27. CT and/or Multimodal MRI exclusion criteria will be: hemispheric strokes < 1.5 cm maximum diameter (on the MRI as seen on the diffusion-weighted imaging or CT)- in order to exclude mild strokes and lacunar strokes of midline shift >1mm or significant hemorrhagic transformation of the acute infarct

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Overall Officials: Dileep Yavagal, MD, Principal Investigator — University of Miami
Locations (1):
- University of Miami Health Systems, Miami, Florida, United States